CLINICAL TRIAL: NCT03968926
Title: Vasoplegia During VA-ECMO for Refractory Cardiogenic Shock : Descriptive Analysis of a Retrospective Cohort
Brief Title: Hypotension During Extracorporeal Circulatory Support Indicated for Cardiogenic Shock
Acronym: RetroECMO-VP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0049
Record Dates: First submitted 2019-05-23; First posted 2019-05-30 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Extracorporeal Life Support; Hypotension; Vasoplegia
Keywords: Cardiogenic shock; Temporary circulatory support; Vasoplegia; Inflammatory response
MeSH Terms: conditions — Hypotension; Vasoplegia; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Plasma: preoperative, ICU admission at POD0 and POD1 samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vasoplegic ECMO: All patients during VA-ECMO support for cardiogenic shock who presented, within 48 hours after implantation, a vasoplegia defined by a norepinephrine dose greater than 0.1µg/kg/min after a 500ml fluid challenge despite overall blood flow (ECMO + native heart) greater than 2l/min/m2 or allowing to achieve 65% of ScvO2
  Interventions: Other: Arterial pressure management during circulatory support by VA-ECMO

INTERVENTIONS:
Other: Arterial pressure management during circulatory support by VA-ECMO — Norepinephrine continuous infusion to maintain mean arterial pressure above 65 mmHg or at a higher level depending of the perfusion pressure targeted for the patient (mean arterial pressure between 65 and 85 mmHg)

SUMMARY:
The cardiogenic shock is characterized by an alteration of organs function following a decrease in cardiac output linked to an impairment of cardiac performance. The prognosis remains poor with mortality between 40 and 50%. Nowadays, Extracorporeal Life Support (ECLS or VA-ECMO) is the referent therapy to restore blood flow in the body when medical treatment is not sufficient. Despite a good blood flow provided by the ECLS, many patients develop a severe hypotension (so called vasoplegia) due to a loss of vascular resistance mainly explained by the inflammatory response to shock and extracorporeal circulation. The treatment of this reaction includes vasopressors (Norepinephrine in usual care) and serum surrogate perfusion to achieve a mean arterial pressure (MAP) above 65 mmHg.

The purpose of this study is to describe the patients with vasoplegia among a retrospective cohort of patients treated with an ECLS in our university center, over the 4 last years, to determine major complication rate (including death, kidney failure and arrythmias) and their outcome. This study will provide consistent data useful for further trials about targets of pressure and treatments to increase blood pressure during ECLS.

DETAILED DESCRIPTION:
Cardiogenic shock is characterized by global tissue hypoperfusion following a decrease in cardiac output by impairing myocardial performance in the absence of hypovolemia. This life-threatening hypoperfusion quickly leads to multiple organs dysfunction with a high risk of cardiac arrest. The main cause is ischemic. The prognosis remains poor with mortality between 40 and 50% and depends on the speed of care by a specialized team. Early etiologic treatment is essential, but initial symptomatic management is based on catecholamines, mainly norepinephrine and dobutamine. The intra-aortic balloon pump showed no improvement in survival in large randomized studies. Refractory cardiogenic shock is defined by the inefficiency or intolerance of catecholamines and the indication of temporary circulatory support should be considered as soon as possible in the absence of contraindications (comorbidities, advanced age, therapeutic limitation). The veno-arterial extracorporeal membrane oxygenation (VA-ECMO or ECLS) is the preferred circulatory assistance in this indication because it provides an overall circulatory support up to 100% of the theoretical cardiac output, with oxygenation, and is quickly implanted peripherally (surgical or percutaneous cannulation of the femoral vein and the femoral artery). However, this extracorporeal circulation also has disadvantages by opposing a major afterload to the failing left ventricle and reducing or even abolishing the pulmonary circulation and blood flow in the heart chambers. In addition, the interaction with the artificial surfaces and the oxygenation membrane of the extracorporeal circuit contributes to the inflammatory response already initiated as a result of low cardiac output, tissue hypoperfusion, mesenteric ischemia and possibly myocardial infarction in case of acute coronary syndrome. This systemic inflammatory response syndrome (SIRS) is similar to sepsis and its main clinical presentation is a vascular dysfunction resulting in vasoplegia and capillary leak syndrome responsible for relative hypovolemia and interstitial inflation.

Since the flow provided by the centrifugal pump is continuous, the blood pressure under VA-ECMO presents low or no pulsatile waves and is better represented by the mean arterial pressure (MAP). The ideal targets of MAP under VA-ECMO are controversial but it is widely accepted that the MAP should not be less than 65mmHg as recommended in septic shock to maintain an acceptable perfusion pressure and should not exceed 95mmHg to limit afterload. Between these limits, the MAP must be individualized according to each situation (hypertensive patient for example). In France, Norepinephrine is the first-line drug to achieve this goal of MAP after correction of volemia, without dose limitation in the absence of currently validated alternative, while resistance mechanisms can be activated, and its efficiency may be limited in case of acidosis. Potential side effects are the occurrence of atrial or ventricular arrhythmias, tachycardia, pro-inflammatory cytokine release, immunosuppression, renal dysfunction.

Management of MAP and vasopressors under VA-ECMO is poorly described in the literature (5), although Norepinephrine is widely used in routine practice. In particular, the investigators do not know the frequency of use and Norepinephrine doses during ECMO-VA, as well as their prognostic involvement. Vasoplegia during VA-ECMO is defined by a Norepinephrine dose greater than 0.1µg/kg/min after a 500ml fluid challenge despite overall blood flow (ECMO + native heart) greater than 2l/min/m2 or allowing to achieve 65% of ScvO2.

This cohort study aims to describe the vasoplegia observed during VA-ECMO, the Norepinephrine treatment characteristics, complications and outcome. The primary end-point is the incidence of a composite criteria of major complications including death, acute kidney injury and arrythmias.

ELIGIBILITY:
Inclusion criteria:

* Refractory cardiogenic shock due to an acute coronary syndrome, a decompensation of chronic heart failure, a infectious or adrenergic myocarditis, or in a post-cardiotomy setting
* Admitted in our intensive care unit between January 2015 and December 2018
* Vasoplegia during the first 48 hours of VA-ECMO requiring more than 0.1µg/kg/min of Norepinephrine continuous infusion

Exclusion criteria:

* Others etiologies of cardiogenic shock : heart transplant dysfunction, right ventricular failure after left ventricular assist device implantation, drug intoxication, hypothermia, pulmonary embolism
* Primary septic shock
* Cardiac arrest with a no-flow time greater than 5 min or a low-flow time greater than 45 min
* Opposition to participate after reception of the information letter

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in intensive care unit for cardiogenic shock at the Montpellier University Hospital and who required a VA-ECMO implantation
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-06-30 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Major complication composite criteria | Up to 7 days for acute kidney injury and arrythmia, and 30 days for death
  Observation of acute kidney injury defined by KDIGO classification 2 or 3, or severe arrythmia (i.e. atrial fibrillation with heart rate above 150bpm or a mean arterial pressure decrease of at least 20%, sustained ventricular tachycardia, ventricular fibrillation), or death

SECONDARY OUTCOMES:
Initial refractory hypotension | Up to 2 hours
  Norepinephrine dose maintained always above 1µg/kg/min during the first 2 hours after VA-ECMO implantation for a minimal mean arterial pressure target at 65mmHg
Refractory vasoplegia | Up to 7 days
  Norepinephrine dose above 1µg/kg/min required to maintain mean arterial pressure above 65mmHg or at the personalized mean arterial pressure target
Mortality rate | Through ICU discharge, an average of 1 month, up to 7, 30 and 90 days
  Overall mortality rate
VA-ECMO free days | At 30 days from the VA-ECMO implantation
  Number of days alive free of VA-ECMO at 30 days after VA-ECMO implantation
Mean arterial pressure | Up to 7 days
  lowest and highest mean arterial pressure (mmHg)
Pulse pressure | Up to 7 days
  lowest and highest pulse pressure (mmHg) defined by the difference between systolic and diastolic pressure
Native cardiac output | Up to 7 days
  lowest and highest cardiac output (L/min) measured by echocardiography (Doppler aortic Velocity Time Integration) or by a pulmonary artery catheter
ECMO flow | Up to 7 days
  lowest and highest flow of VA-ECMO (L/min)
Lactate | Up to 7 days
  Highest lactate level of the day (mmol/l)
ScvO2 | Up to 7 days
  Highest and lowest central venous oxygen saturation (%)
Urine output | Up to 7 days
  Total urine output of the day (ml/24H)
Hydric balance | Up to 7 days
  Total hydric balance calculated from day 0 to day 7 (ml)
Hospital stay | through study completion, an average of 3 month
  Length (days) of hospital stay from the VA-ECMO implantation before current care ward discharge (excluding rehabilitation time)
Intensive care unit stay | through study completion, an average of 3 month
  Length (days) of intensive care unit stay from the VA-ECMO implantation
Issue of VA-ECMO | 7 days after VA-ECMO withdrawal
  Status after VA-ECMO including death, heart transplant, ventricular assist device, recovery, shock recurrence, therapy limitation
Serious adverse events | Trough VA-ECMO time completion, an average of 2 weeks
  Stroke, bleeding requiring blood transfusion or surgical revision, limb ischemia, mesenteric ischemia, documented infection
Organ failure assessment | At day 0, 5 and 10 after VA-ECMO implantation
  Sequential Organ Failure Assessment score (0 to 24), higher values represent a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Gaudard, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Diepen S, Katz JN, Albert NM, Henry TD, Jacobs AK, Kapur NK, Kilic A, Menon V, Ohman EM, Sweitzer NK, Thiele H, Washam JB, Cohen MG; American Heart Association Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Quality of Care and Outcomes Research; and Mission: Lifeline. Contemporary Management of Cardiogenic Shock: A Scientific Statement From the American Heart Association. Circulation. 2017 Oct 17;136(16):e232-e268. doi: 10.1161/CIR.0000000000000525. Epub 2017 Sep 18. PMID 28923988
- [Background] Tanaka D, Shimada S, Mullin M, Kreitler K, Cavarocchi N, Hirose H. What Is the Optimal Blood Pressure on Veno-Arterial Extracorporeal Membrane Oxygenation? Impact of Mean Arterial Pressure on Survival. ASAIO J. 2019 May/Jun;65(4):336-341. doi: 10.1097/MAT.0000000000000824. PMID 29762229